CLINICAL TRIAL: NCT00609310
Title: Dietary Supplementation With Bioflavonoids for the Prevention of the Recurrence of Neoplasia in Patients With Resected Colorectal Carcinoma
Brief Title: Dietary Bioflavonoid Supplementation for the Prevention of Neoplasia Recurrence
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Flav-Hoe-CCR
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer
Keywords: clinical trial; flavonoid treatment; neoplasia recurrence; colorectal cancer; polypectomy; adenoma in Colon; Neoplasia Recurrence Rates; postpolypectomy patients
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Flavonoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Flavonoid treatment
  Interventions: Dietary Supplement: Flavonoids

INTERVENTIONS:
Dietary Supplement: Flavonoids — Nutritional Supplement: flavonoid mixture with 20 mg apigenin and 20 mg epigallocathechin gallate as tablets per day

SUMMARY:
Prove the hypothesis that dietary supplementation with bioflavonoids will diminish the recurrence rate of colonic neoplasia, we will implement a clinical trial comparing bioflavonoids and placebo in a double blind randomized clinical trial. To use a standardised supplementation of bioflavonoids, a commercially available preparation (Flavo-Natin®) will be used.

DETAILED DESCRIPTION:
The preparation contains a mixture of 200mg chamomile and tea (green tea) extract which contains naturally occurring bioflavonoids (2%) together with vitamins and folic acid. This flavonoids mixture will be applied for 3 years and the compliance and effects of this treatment will be determined by measuring the serum concentrations of apigenin and EGCG of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had a recent surgical resection of colorectal cancer with pathologically proven stage 2 or stage 3 (without adjuvant chemotherapy or after completion of adjuvant chemotherapy) according to UICC. The time interval for recruitment should be within 3-12 month after surgery.
* Male or female
* caucasian
* 50 to 75 years old
* Broca-index: between -20 and +25%
* who are willing and capable to confirm written consent to enrolment after ample information has been provided
* who are in a stable condition that it can be expected that no changes in relevant medical conditions will occur during the study

Exclusion Criteria:

* subjects with any major relevant clinical abnormality (as based on extensive medical history, physi-cal examination, vital signs)
* subjects with active cancer
* subjects with any major clinically relevant laboratory abnormality.
* subjects who participated in another trial with any investigational substance within the last 4 weeks
* subjects who are known or suspected to be (social) drug dependent, incl. those drinking more than moderately and who are not willing to abstain from alcohol abuse during the active study phase
* subjects who adhere to a extreme diet or lifestyle that might interfere with the investigation
* subjects who are known or suspected not to comply with the study directives and/or who are known or suspected not to be reliable or trustworthy
* subjects who are known or suspected not to be capable of understanding and evaluating the in-formation that is given to them as part of the formal information policy (informed consent), in par-ticular regarding the risks and discomfort to which they would agree to be exposed

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of neoplasia | 3 years

SECONDARY OUTCOMES:
Recurrence free survival, Overall survival, Serum-Flavonoid levels of patients | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Harald Hoensch, Professor, Study Chair — Community Hospital Darmstadt, Germany
Locations (1):
- community Hospital, Darmstadt, Hesse, Germany